CLINICAL TRIAL: NCT04731727
Title: Safety and Effectiveness of the CCL Vario System for Corneal Collagen Cross-Linking in Eyes With Corneal Thinning Conditions
Brief Title: Treating Corneal Thinning Conditions With CCL Vario Riboflavin (CXL)
Acronym: CXL
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kent Wellish MD (Other)
Responsible Party: Sponsor-Investigator, Kent Wellish MD, President and Medical Director, Wellish Vision Institute
Organization: Wellish Vision Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0000
Record Dates: First submitted 2021-01-21; First posted 2021-02-01 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Keratoconus, Unstable
MeSH Terms: conditions — Keratoconus | interventions — Riboflavin; Ultraviolet Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cross linking treatment for corneal thinning (Experimental): Cornea will be saturated with Vitamin B2 (Riboflavin) and then treated with 365 nm wavelength ultra violet light.
  Interventions: Drug: Riboflavin

INTERVENTIONS:
Drug: Riboflavin — Corneal cross linking achieved by combination of Riboflavin and ultraviolet light
  Other Names: Ultra violet light

SUMMARY:
Study is testing the efficacy of treating corneal thinning conditions with Vitamin B2 (Riboflavin) and the application on UV Light.

DETAILED DESCRIPTION:
Corneal thinning conditions, i.e. keratoconus or ectasia, weaken the cornea which then causes the front of the eye to bulge out. This results in distorted vision and could eventually result in the need for a cornea transplant. This study proposes to conclude that saturating the cornea with vitamin B2 (Riboflavin) and then applying 365nm wavelength of Ultra Violet Light will result in the various layers of corneal tissue linking together. This cross linking results in a stronger cornea which is designed to halt the progression of keratoconus or ectasia. This treatment is already being successfully used in Europe.

ELIGIBILITY:
Inclusion Criteria:

* Presence of central or inferior corneal steepening
* Axial topography consistent with keratoconus, post-surgical ectasia, or pellucid marginal degeneration
* Presence of one or more findings associated with keratoconus or pellucid marginal degeneration, such as:
* Fleischer ring
* Vogt's striae
* Decentered corneal apex
* Munson's sign
* Rizutti's sign
* Apical corneal scarring consistent with Bowman's breaks
* Scissoring of the retinoscopic reflex
* Crab-claw appearance on topography
* Steepest keratometry (Kmax) value > or = 47.20 D
* I-S keratometry difference > 1.5 D on the Orbscan map
* Posterior corneal elevation > 16 microns
* Thinnest corneal point < 485 microns
* Post LASIK/PRK stromal ablation depth < 300 microns or expected keratometry > 47.2 D, or post-PRK/SMILE in keratoconus suspect eyes
* Bacterial or fungal corneal keratitis persistent and not responding despite > 2 weeks of standard antimicrobial therapy or with rapid progression of corneal thinning, with loss of > 25% corneal thickness
* Contact Lens Wearers Only:
* Removal of contact lenses for the required period of time prior to the screening refraction:

Contact Lens Type Minimum Discontinuation Time Soft 1 Week Soft Extended Wear 2 Weeks Soft Toric 3 Weeks Rigid Gas Permeable 2 Weeks per decade of wear

* Signed written informed consent
* Willingness and ability to comply with schedule for follow-up visits

Exclusion Criteria:

* Eyes classified as either normal or atypical normal on the severity grading scheme
* Corneal pachymetry at the screening exam that is < 400 microns at the thinnest point in the eye(s) to be treated when the transepithelial (isotonic) riboflavin solution alone will be used or < 300 microns when the hypotonic riboflavin will be used.
* Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications, for example:

  1. History of or active corneal disease (e.g., herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, acanthamoeba, etc.)
  2. Clinically significant corneal scarring in the CXL treatment zone that is not related to keratoconus or, in the investigator's opinion, will interfere with the cross linking procedure
* Pregnancy (including plan to become pregnant) or lactation during the course of the study
* A known sensitivity to study medications
* Patients with nystagmus or any other condition that would prevent a steady gaze during the CXL treatment or other diagnostic tests
* Patients with a current condition that, in the physician's opinion, would interfere with or prolong epithelial healing

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Best Corrected Visual Acuity | Baseline and 1 year
  Use a standard eye chart to determine changes in the subject's best Visual Acuity (with glasses or contact) performed by research staff
Change in Uncorrected Visual Acuity | Baseline and 1 year
  Use a standard eye chart to determine changes in the subject's best Visual Acuity (without glasses or contact) performed by clinic technician
Occurrence of Adverse Events | Through study completion, an average of 1 year
  Surgeon notes any occurrence of adverse events related to the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kent L Wellish, MD, Principal Investigator — Wellish Vision Institute

IPD SHARING:
Plan to Share IPD: No
Unidentifiable patient data and pre- and post-op results will be shared.